CLINICAL TRIAL: NCT00163514
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Clinical Trial Designed to Assess the Efficacy and Safety of Ciclesonide Applied as a Nasal Spray at Three Dose Levels (200 Mcg, 100 Mcg, or 25 Mcg, Once Daily) in the Treatment of Perennial Allergic Rhinitis (PAR) in Patients 6-11 Years of Age
Brief Title: Safety and Effectiveness of Ciclesonide Nasal Spray in Children (6 to 11 Years) With Perennial Allergic Rhinitis (BY9010/M1-403)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BY9010/M1-403
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Perennial Allergic Rhinitis; Allergic Rhinitis; Hay Fever
Keywords: Allergy; Perennial Allergic Rhinitis; Allergic Rhinitis; Hay Fever
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Hypersensitivity | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of ciclesonide nasal spray as compared with placebo (inactive substance) nasal spray in relieving symptoms of perennial allergic rhinitis.

ELIGIBILITY:
Main Inclusion Criteria:

* General good health, other than perennial allergic rhinitis
* History and diagnosis of perennial allergic rhinitis by skin prick test
* Parent/caregiver must be capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent and comply with all study requirements (visits, record-keeping, etc.)

Main Exclusion Criteria:

* Participation in any investigational drug trial within the 30 days preceding the Screening Visit or at any time during the trial
* Use of any prohibited concomitant medications as defined by the study protocol
* Non-vaccinated exposure to, or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 636
Dates: Start 2004-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
changes in Total Nasal Symptom Score

SECONDARY OUTCOMES:
safety, changes in symptoms

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (71):
- United States (55):
  - Altana Pharma/Nycomed, Oxford, Alabama
  - Altana Pharma/Nycomed, Huntington Beach, California
  - Altana Pharma/Nycomed, Mission Viejo, California
  - Altana Pharma/Nycomed, Newport Beach, California
  - Altana Pharma/Nycomed, Orange, California
  - Altana Pharma/Nycomed, Palmdale, California
  - Altana Pharma/Nycomed, San Diego, California
  - Altana Pharma/Nycomed, San Jose, California
  - Altana Pharma/Nycomed, Stockton, California
  - Altana Pharma/Nycomed, Walnut Creek, CA, California
  - Altana Pharma/Nycomed, Coral Gables, Florida
  - Altana Pharma/Nycomed, Ocala, Florida
  - Altana Pharma/Nycomed, Atlanta, Georgia
  - Altana Pharma/Nycomed, Gainesville, Georgia
  - Altana Pharma/Nycomed, Savannah, Georgia
  - Altana Pharma/Nycomed, Normal, Illinois
  - Altana Pharma/Nycomed, Indianapolis, Indiana
  - Altana Pharma/Nycomed, Dubuque, Iowa
  - Altana Pharma/Nycomed, Overland Park, Kansas
  - Altana Pharma/Nycomed, Metairie, Louisiana
  - Altana Pharma/Nycomed, Shreveport, Louisiana
  - Altana Pharma/Nycomed, Rockville, Maryland
  - Altana Pharma/Nycomed, Wheaton, Maryland
  - Altana Pharma/Nycomed, North Dartmouth, Massachusetts
  - Altana Pharma/Nycomed, Minneapolis, Minnesota
  - Altana Pharma/Nycomed, Jefferson City, Missouri
  - Altana Pharma/Nycomed, Rolla, Mo, Missouri
  - Altana Pharma/Nycomed, St Louis, Missouri
  - Altana Pharma/Nycomed, Papillion, Nebraska
  - Altana Pharma/Nycomed, Brick, New Jersey
  - Altana Pharma/Nycomed, Skillman, New Jersey
  - Altana Pharma/Nycomed, Liverpool, New York
  - Altana Pharma/Nycomed, Raleigh, North Carolina
  - Altana Pharma/Nycomed, Canton, Ohio
  - Altana Pharma/Nycomed, Cincinnati, OH, Ohio
  - Altana Pharma/Nycomed, Sylvania, Ohio
  - Altana Pharma/Nycomed, Medford, Oregon
  - Altana Pharma/Nycomed, Portland, Oregon
  - Altana Pharma/Nycomed, Easton, Pennsylvania
  - Altana Pharma/Nycomed, Hershey, Pennsylvania
  - Altana Pharma/Nycomed, Upland, Pennsylvania
  - Altana Pharma/Nycomed, Charleston, South Carolina
  - Altana Pharma/Nycomed, Moncks Corner, South Carolina
  - Altana Pharma/Nycomed, Spartanburg, South Carolina
  - Altana Pharma/Nycomed, Austin, Texas
  - Altana Pharma/Nycomed, El Paso, Texas
  - Altana Pharma/Nycomed, Fort Worth, Texas
  - Altana Pharma/Nycomed, Friendswood, Texas
  - Altana Pharma/Nycomed, Houston, Texas
  - Altana Pharma/Nycomed, Katy, Texas
  - Altana Pharma/Nycomed, Salt Lake City, Utah
  - Altana Pharma/Nycomed, South Burlington, Vermont
  - Altana Pharma/Nycomed, Burke, Virginia
  - Altana Pharma/Nycomed, Richmond, Virginia
  - Altana Pharma/Nycomed, Spokane, Washington
- Canada (16):
  - Altana Pharma/Nycomed, Hamilton
  - Altana Pharma/Nycomed, Hamilton, on
  - Altana Pharma/Nycomed, Kanata, on
  - Altana Pharma/Nycomed, London
  - Altana Pharma/Nycomed, London,ON
  - Altana Pharma/Nycomed, Mississauga
  - Altana Pharma/Nycomed, Montreal, QC
  - Altana Pharma/Nycomed, Niagara Falls
  - Altana Pharma/Nycomed, Oshawa, on
  - Altana Pharma/Nycomed, Ottawa
  - Altana Pharma/Nycomed, Ottawa, on
  - Altana Pharma/Nycomed, Saskatoon,SK
  - Altana Pharma/Nycomed, Ste-Foy PQ
  - Altana Pharma/Nycomed, Toronto
  - Altana Pharma/Nycomed, Toronto, on
  - Altana Pharma/Nycomed, Winnipeg

REFERENCES:
- See also: BY9010-M1-403-RDS-2005-12-09.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4531&filename=BY9010-M1-403-RDS-2005-12-09.pdf